CLINICAL TRIAL: NCT00351208
Title: The Efficacy of Spinal Cord Stimulation at Varying Stimulation Frequencies and Pulse-Widths
Brief Title: Spinal Cord Stimulation Efficacy Measures
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Neurosurgery & Neuroscience Associates, PLLC (Other)
Collaborators: MedtronicNeuro (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-20-
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2006-07-12 (Estimated); Status verified 2006-06

CONDITIONS: Chronic Pain in the Trunk and Limbs
Keywords: Spinal cord stimulation; Spinal cord stimulation efficacy; Spinal cord stimulators; Stimulation frequencies; Stimulation pulse-widths; Varying settings

INTERVENTIONS:
Device: Medtronic Manufactured Spinal Cord Stimulators

SUMMARY:
The purpose of the study is to measure the efficacy of varying spinal cord stimulation frequencies and pulse-width settings on chronic pain management. The spinal cord stimulator settings that are most effective in chronic pain management hope to be revealed for the purposes of this study. In this double-blind study, both the patient and the staff will not be aware of the spinal cord stimulator settings for each patient each week. The representative that will set the settings each week will be blinded to the identity of each patient and will set the spinal cord stimulator from another room. While there are few papers that show the efficacy of spinal cord stimulation in treating chronic pain, there has yet to be a study performed that measures the role of stimulation frequency and pulse-widths. This study hopes to be the first.

DETAILED DESCRIPTION:
For a total of 9 weeks, patients will be randomized to 9 stimulation frequency and pulse-width setting combinations. The patient will stay with these settings for a week at a time. Prior to the patient's first office visit, he/she will be asked to take a chest x-ray. The patient will also repeat this chest x-ray at the end of the study. Each patient will be asked to provide daily information regarding pain medication usage, spinal cord stimulation usage, amplitude settings, and pain ratings. Additionally, patients will fill out the Multidimensional Pain Inventory (MPI) and the McGill Pain Questionnaire (MPQ) every Monday when they come to the office, before he/she is randomized to the new settings for the week. The patient will also receive a call from the research assistant to see how he/she is doing that week and the patient will be provided with all the pertinent contact information to call at any time to ask questions. The patient can withdraw from the study completely at any point or drop out of the settings for the week. The patient will have a follow-up visit a month from the study's end date to discuss how the patient has been managing his/her pain at his/her spinal cord stimulator settings. Each patient will be compensated for completing the study. Efficacy will be measured based on the patient's answers to the pain probes, device usage, and medication usage.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have SCS implanted for at least 2 months before study start date
* The patient must be at least 18 years old
* The patient must currently be receiving pain relief from SCS usage
* The patient must be willing to participate in a 9-week study
* The patient must have at least 20% of battery life remaining in his/her spinal cord stimulator
* The patient must be able to tolerate Vicodin-Extra Strength as well as Tylenol, but can also take their own pain medication if it is not one of the two mentioned

Exclusion Criteria:

* The patient is pregnant or intends to become pregnant during the course of the study.
* The patient by report, and/or by physician assessment, exhibits any or all of the following, which might bias reporting of treatment outcome:

A strong untreated dependency on prescription medication such as benzodiazepines and narcotic analgesics.

A strong potential for secondary gain issues.

A significant, untreated psychiatric comorbidity.

* The patient possesses a coexisting clinically relevant or disabling chronic pain problem not treated by SCS
* The patient has been diagnosed with unstable angina
* The patient receives a Karnofsky's performance score of <60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-05; Study Completion 2006-08

PRIMARY OUTCOMES:
Percent pain relief obtained during the one-month follow-up compared to baseline
The magnitude of change in other indexes of function, such as MPI, during the one-month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Louis G Cornacchia, MD, Principal Investigator — New York Neurosurgery & Neuroscience Associates, PLLC
Locations (2):
- United States (2):
  - The Brookdale University Hospital and Medical Center, Brooklyn, New York
  - New York Neurosurgery & Neuroscience Associates, PLLC, Rockville Centre, New York

REFERENCES:
- [Background] Mailis-Gagnon A, Furlan AD, Sandoval JA, Taylor R. Spinal cord stimulation for chronic pain. Cochrane Database Syst Rev. 2004;(3):CD003783. doi: 10.1002/14651858.CD003783.pub2. PMID 15266501
- [Background] Barbetakis N, Antoniadis T, Tsilikas C. Results of chemical pleurodesis with mitoxantrone in malignant pleural effusion from breast cancer. World J Surg Oncol. 2004 May 20;2:16. doi: 10.1186/1477-7819-2-16. PMID 15153245
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473